CLINICAL TRIAL: NCT05828446
Title: Prospective Comparison of Diagnostic Performance and Cost-effectiveness of US and Abbreviated MRI for Hepatocellular Carcinoma Screening
Brief Title: Improving Hepatocellular Carcinoma Screening
Acronym: AMRIK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Naik Vietti Violi (Other)
Responsible Party: Sponsor-Investigator, Naik Vietti Violi, Radiologist, Principal investigator, University of Lausanne Hospitals
Organization: University of Lausanne Hospitals (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CER-VD 2022-D0116
Record Dates: First submitted 2023-01-19; First posted 2023-04-25 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Magnetic Resonance Imaging; Hepatocellular Carcinoma; Screening; Contrast-enhanced US
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Intervention Model Description: single center interventional prospective study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HCC screening population according to European Association for the Study of the Liver recommendation (Experimental)
  Interventions: Device: MRI

INTERVENTIONS:
Device: MRI — To compare the diagnostic performance of US+/- Constrast-enhanced US and AMRI for HCC detection in an at-risk population
  Other Names: Constrast-enhanced US

SUMMARY:
This is a monocentric, single blind, interventional, single arm study. It is designed to compare the rates of detection of hepatocellular carcinoma (HCC) by ultrasound (US) used in clinical routine vs. abbreviated magnetic resonance imaging (AMRI). The hypothesis is that dynamic AMRI with extracellular contrast agent injection has a higher patient-level detection rate of HCC than screening US and non-contrast AMRI.

Interested and eligible patients will be enrolled and undergo HCC screening rounds including US +/- contrast-enhanced US (clinical routine) and screening MRI within the same week bi-annually.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients with chronic liver disease and indication for HCC screening according to the European Association for the Study of the Liver recommendations.
* Informed Consent signed by the subject

Exclusion Criteria:

* History of HCC
* History of other malignancy
* Prior liver nodule categorized as LI-RAD 4, 5 or M
* History of liver transplantation
* Pregnancy
* MRI or MRI contrast agent precaution
* Any other condition making the patient unsuitable for the study
* Patient's refusal of transmission of relevant medical conditions found on the medical examinations performed during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
To compare the diagnostic performance of US+/- CEUS and AMRI for HCC detection in an at-risk population | Through study completion, an average of 1 year.
  The patients will undergo all the normal follow-up according to clinical recommendations, consisting of a bi-annual clinical visit in the gastro-enterology department and an US. The US will be followed by CEUS in case of suspicious lesion. On the same week, the study participants will undertake MRI.
  The data of the full MRI will be used to reconstruct two different AMRI sets for reading: non-contrast (NC-) and dynamic (Dyn-) AMRI.
  The endpoint is the rate of HCC detection. Outcome measures will be compared in terms of ROC curve and AUC.

SECONDARY OUTCOMES:
Compare the patient-level accuracy, sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV) of US +/- CEUS vs. AMRI for HCC. | Through study completion, an average of 1 year.
  Diagnostic performance of the different tests [(1)US alone, (2) US + CEUS, (3) NC-AMRI, (4) Dyn-AMRI] will be compared using all patient information (including complete MRI and pathology) as the reference standard.
  Outcome measures will be compared in terms accuracy, sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV)
Evaluate patient satisfaction and comfort with US +/- CEUS vs. AMRI with a questionnaire | Once, after the first screening round (US+/-CEUS and MRI), 6 months
  In order to evaluation patient's opinion a survey regarding patient experience and opinion to the different test will be performed.
  Outcome will be measured in term of level of confort using a 5-scale score: from low discomfort to high discomfort:
  1. No discomfort
  2. Low discomfort
  3. Neutral
  4. Comfort
  5. high comfort
To develop and test a DL model for HCC detection based on AMRI. | Through study completion, an average of 1 year.
  AMRI DL based model will be analysed in terms of (1) diagnostic performance (ROC, AUC, sensitivitiy, specificity, accuracy) and (2) time savings compared to AMRI read by a radiologist.
To perform a cost-effectiveness analysis comparing US to different alternative screening strategies for HCC in Switzerland. | Through study completion, an average of 1 year.
  Cost effectiveness analysis will be perfomed by building a model using all study data: patient characteristics, exam diagnostic performance and patient management costs.
  Outcome will be analysed in terms of Lifetime costs, quality adjusted life expectancy
To perform a cost-effectiveness analysis comparing US to different alternative screening strategies for HCC in Switzerland. | Through study completion, an average of 1 year.
  Cost effectiveness analysis will be perfomed by building a model using all study data: patient characteristics, exam diagnostic performance and patient management costs.
  Outcome will be analysed in terms of incremental costs effectiveness ratios.

CONTACTS AND LOCATIONS:
Overall Officials: Naik Vietti Violi, MD, Principal Investigator — University of Lausanne Hospitals
Locations (1):
- Lausanne University Hospital, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided